CLINICAL TRIAL: NCT03890445
Title: GIANT - A Multicenter, Prospective, Observational Study of Real-world Anti-TNFa Treatment Regimens of Hyrimoz™ (Adalimumab Biosimilar) or Zessly™ (Infliximab Biosimilar) in Patients With Crohn's Disease
Brief Title: Real-world Study of Anti-TNFa Treatment Regimes of Hyrimoz or Zessly in Patients With Crohn´s Disease
Acronym: GIANT
Status: Completed | Type: Observational
Sponsor: Sandoz (Industry)
Responsible Party: Sponsor
Other Study IDs: CGPN017A2001; NCT03930030 (obsolete NCT alias); NCT04022083 (obsolete NCT alias)
Record Dates: First submitted 2019-03-22; First posted 2019-03-26 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Crohn´s Disease
Keywords: Crohn´s Disease; Inflammatory Bowel Disease; Adalimumab; Infliximab; Biosimilar; IBD-Index
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Adalimumab Biosimilar (Hyrimoz): Patients with moderate-to-severe CD receiving Hyrimoz™ treatment according to the Hyrimoz™ label at the discretion of the investigator
- Infliximab Biosimilar (Zessly): Patients with moderate-to-severe CD receiving Zessly™ treatment according to the Zessly™ label at the discretion of the investigator

SUMMARY:
Hyrimoz™ was developed as a biosimilar to HumiraTM (INN: adalimumab) and Zessly™ was developed as a biosimilar to RemicadeTM (INN: infliximab). Within the Biosimilar Development Program of Hyrimoz™ and Zessly™, two clinical confirmatory efficacy and safety studies were conducted: Hyrimoz™ in plaque psoriasis and Zessly™ in rheumatoid arthritis. Both confirmatory Phase III studies demonstrated equivalent efficacy and similar safety and immunogenicity of Hyrimoz™ to HumiraTM and Zessly™ to RemicadeTM, respectively.

The current study is designed to provide a systematic and consistent overview of the real-world data in biologic-naïve patients with moderate-to-severe Crohn's disease (CD). The data collected in this observational trial will be used to increase the knowledge of the effectiveness of Hyrimoz™ and Zessly™ in clinical routine care in patients with moderate-to-severe CD.

ELIGIBILITY:
The inclusion and exclusion criteria are to ensure the enrollment of patients receiving the drug according to the label of Hyrimoz™ and the label of Zessly™. Patients observed in this study need to meet all of the following inclusion criteria and none of the exclusion criteria at enrollment:

Inclusion criteria

1. Confirmed diagnosis of CD
2. Harvey-Bradshaw Index (HBI) ≥ 5
3. Treatment failure upon steroids / topical budesonide with or without immunosuppressants
4. Males and females ≥ 18 years of age at enrollment
5. Biologic-naive patients scheduled to receive Hyrimoz™ or Zessly™ and patients already receiving Hyrimoz™ or Zessly™ according to the label and at the discretion of the investigator for up to three months prior enrollment
6. Provision of signed informed consent form

Exclusion criteria

1. Patients with CD in clinical remission (HBI < 5)
2. Hemoglobin < 8.5 g/dL
3. Patients at imminent risk of scheduled intestinal surgery (stenosis, strictures, internal fistula)
4. Any contraindications to Hyrimoz™ or Zessly™ according to the prescribing recommendations in each country
5. Participation in an interventional clinical trial for immune-mediated inflammatory diseases (IMIDs) or having received any investigational agent or procedure within 30 days prior to enrollment (consenting)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It is planned to enroll a total of 1,600 patients.
  The following patient groups will be observed:
  * Patients with moderate-to-severe CD receiving Hyrimoz™ treatment according to the Hyrimoz™ label at the discretion of the investigator
  * Patients with moderate-to-severe CD receiving Zessly™ treatment according to the Zessly™ label at the discretion of the investigator
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2020-05-08 (Actual); Study Completion 2020-05-08 (Actual)

PRIMARY OUTCOMES:
The proportion of patients in corticosteroid-free remission defined as HBI (Harvey-Bradshow Index) ≤ 4 at Week 52 | week 52
  This is a prospective, observational study that does not impose a therapy protocol, diagnostic or therapeutic procedure, or a visit schedule. Patients will be treated according to the local prescribing information, and routine medical practice in terms of visit frequency and types of assessments performed; only these data will be collected as part of the study.

SECONDARY OUTCOMES:
Time to progression of a composite endpoint | 6 years
  Composite endpoint defined as the occurrence of one of the following events :
  * Disease-related surgery, or
  * Disease-related hospital admission for > 3 days (including treatment-related side effects), or
  * Serious disease-related complications
Incidence of adverse events | 6 years
  • Incidence of Adverse Events (AE) in patients receiving Hyrimoz™ or Zessly™
Measurement of the Inflamatory Bowel Disease (IBD) index over an observation period | 4 years
Assessing correlation of the diagnostic and treatment-monitoring procedures (imaging procedures and disease-related laboratory parameters) in patients receiving Hyrimoz™ or Zessly™ over an observation period | 4 years
Assessing QoL (Quality of Life scale) of patients receiving Hyrimoz™ or Zessly™ over an observation period | 4 years
Therapy persistence and treatment adherence (measured by the number of dose interruptions of Hyrimoz™ or Zessly™ without drug holidays more than 4 months). | 4 years
  Observational study

CONTACTS AND LOCATIONS:
Locations (18):
- Austria (3):
  - Sandoz Investigational Site, Innsbruck
  - Sandoz Investigational Site, Salzburg
  - Sandoz Investigational Site, Vienna
- Germany (10):
  - Sandoz Investigational Site, Herne, North Rhine-Westphalia
  - Sandoz Investigational Site, Altenholz
  - Sandoz Investigational Site, Alzey
  - Sandoz Investigational Site, Berlin
  - Sandoz Investigational Site, Dachau
  - Sandoz Investigational Site, Iserlohn
  - Sandoz Investigational Site, Jerichow
  - Sandoz Investigational Site, Munich
  - Sandoz Investigational Site, Münster
  - Sandoz Investigational Site, Saarbrücken
- Poland (2):
  - Sandoz Investigational Site, Piotrkow Trybunalski
  - Sandoz Investigational Site, Włocławek
- Spain (2):
  - Sandoz Investigational Site, Ferrol
  - Sandoz Investigational Site, Madrid
- Sandoz Investigational Site, Örebro, Sweden

REFERENCES:
- See also: Study Results — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17835